CLINICAL TRIAL: NCT06566079
Title: A Phase 1, Open-Label, Multicenter, FIH Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Preliminary Efficacy of ISM6331 in Participants With Advanced/Metastatic Malignant Mesothelioma or Other Solid Tumors
Brief Title: Study of ISM6331 in Participants With Advanced/Metastatic Malignant Mesothelioma or Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISM6331-101
Record Dates: First submitted 2024-08-13; First posted 2024-08-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Malignant Mesothelioma; Metastatic Malignant Solid Tumor; Advanced Solid Tumor
Keywords: Transcriptional enhanced associate domain (TEAD); TEAD inhibitor; ISM6331; Hippo pathway; YAP/TAZ-TEAD
MeSH Terms: conditions — Mesothelioma, Malignant; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): Patients will receive ISM6331 once daily in sequential cohorts of increasing doses.
  Interventions: Drug: ISM6331
- Part 2 Dose Selection Optimization (Experimental): Participants will receive ISM6331 once daily at each dose level from the two dose levels recommended by Study Review Committee.
  Interventions: Drug: ISM6331

INTERVENTIONS:
Drug: ISM6331 — Dosage form: Capsule for oral administration.
  Frequency of administration: Once daily overall of treatment.

SUMMARY:
This is a Phase 1, open-label, multicenter, FIH study to evaluate the safety, tolerability, recommended Phase 2 dose (RP2D), PK/PD, and preliminary anti-tumor activity of ISM6331 in participants with advanced or metastatic malignant mesothelioma or other solid tumors. The study consists of two parts, a dose escalation part (Part 1) and a dose selection optimization part (Part 2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with age ≥18 years at the time of signing the informed consent.
2. Histologically confirmed unresectable advanced or metastatic malignant mesothelioma or other solid tumors, who have failed standard therapy or for whom no effective standard therapy exists, participants for part 1 is regardless of the presence or absence of the genetic alterations of the Hippo pathway, but for part 2 participants with solid tumors other than mesothelioma, genetic testing documentation must demonstrate Hippo signaling pathway dysregulation.
3. Participants with malignant mesothelioma must have prior exposure to at least immune checkpoint therapy and platinum-based chemotherapy.
4. Presence of at least one evaluable lesion in Part 1 or one measurable target lesion in Part 2 according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) for participants with non-pleural mesothelioma or other solid tumors and modified RECIST (mRECIST) v1.1 for participants with malignant pleural mesothelioma.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1.
6. Life expectancy of ≥12 weeks as judged by the investigator.
7. Adequate organ function as determined by medical assessment (within 7 days prior to the first dose of study treatment).
8. Capable of providing signed informed consent form (ICF) and complying with the requirements and restrictions listed in the ICF and in this study protocol.

Exclusion Criteria:

1. Participants who have previously received a TEAD inhibitor.
2. Participation in other therapeutic clinical studies within 28 days or 5 half-lives (whichever is shorter) prior to first dose of study treatment.
3. Anti-tumor therapy within 28 days or 5 half-lives (whichever is shorter) prior to first dose of study treatment.
4. Known active central nervous system (CNS) primary tumor or untreated CNS metastases.
5. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases.
6. Unwillingness or unable to comply with the requirements of oral drug administration, or presence of a gastro-intestinal condition
7. Have prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, laboratory abnormality or any other conditions that, in the investigator's opinion, would not be in the best interest of the participant; or that could alter the absorption, distribution, metabolism, or excretion of the study treatment; or impair the assessment of study result.
8. Currently receiving any of Strong inhibitors or inducers of P-gp, or Sensitive substrates of P-gp, CYP1A2, CYP2B6, and CYP3A4 that cannot be discontinued 14 days or 5 half-lives for inhibitors or substrates (whichever is shorter) prior to the first dose of study treatment.

Other protocol inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT). | Day 1 up to Day 31
  DLT is defined as any adverse event which meets DLT criteria unless it is clearly related to disease progression or intercurrent illness during the first 31 days after the initiation of treatment in the dose escalation part (Part 1).
Incidence and severity of adverse events (AEs) | Approximately 12 months.
  Adverse events are assessed based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 [NCI CTCAE v5.0]
Incidence of clinically significant abnormalities in laboratory values, vital signs, physical examination, and electrocardiogram (ECG) measurements. | Approximately 12 months.
  Regular monitoring and assessment of vital signs (pulse rate, blood pressure, respiratory rate, and temperature), physical examinations, laboratory values, ECG, and other safety examinations by investigators.
Recommended Phase 2 Dose (RP2D) | Approximately 40 months
  The RP2D will be recommended by safety review committee (SRC) upon reviewing all available safety, tolerability, pharmacokinetics/pharmacodynamics, and preliminary efficacy data from Part 1 and Part 2.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Approximately 12 months
  Pharmacokinetics (PK) parameters of ISM6331 after dose of ISM6331 will be assessed.
Area under the concentration-time curve (AUC) | Approximately 12 months
  Pharmacokinetics (PK) parameters of ISM6331 after dose of ISM6331 will be assessed.
Terminal half-life (t1/2) | Approximately 12 months
  Pharmacokinetics (PK) parameters of ISM6331 after dose of ISM6331 will be assessed.
Objective response rate (ORR). | Approximately 12 months
  Efficacy assessments will be conducted at baseline and every 8 weeks within the first 6 months after the first dose of study treatment, then every 12 weeks thereafter, until progressive disease confirmed by the investigator, start of a new anti-tumor treatment, death, lost to follow-up, or withdrawal from the study, whichever occurs first.
Best objective response (BOR). | Approximately 12 months
  Efficacy assessments will be conducted at baseline and every 8 weeks within the first 6 months after the first dose of study treatment, then every 12 weeks thereafter, until progressive disease confirmed by the investigator, start of a new anti-tumor treatment, death, lost to follow-up, or withdrawal from the study, whichever occurs first.
Duration of response (DoR). | Approximately 12 months
  Efficacy assessments will be conducted at baseline and every 8 weeks within the first 6 months after the first dose of study treatment, then every 12 weeks thereafter, until progressive disease confirmed by the investigator, start of a new anti-tumor treatment, death, lost to follow-up, or withdrawal from the study, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - The University of Chicago Medical Center - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Oncology - Austin, Austin, Texas
- China (3):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Sun Yat-Sen University Cancer Center, Guangzhou